CLINICAL TRIAL: NCT00219375
Title: Efficacy and Safety of Sivelestat Sodium Hydrate in Acute Lung Injury Associated With Systemic Inflammatory Response Syndrome, Compared With the Conventional Treatment in Japan
Brief Title: Study of Sivelestat Sodium Hydrate in Acute Lung Injury (ALI) Associated With Systemic Inflammatory Response Syndrome (SIRS) in Japan
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-601/602/603-0001
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2012-06

CONDITIONS: Acute Lung Injury; Systemic Inflammatory Response Syndrome
Keywords: sivelestat sodium hydrate; acute lung injury; systemic inflammatory response syndrome; Elaspol; Acute Lung Injury (ALI) Associated With Systemic Inflammatory Response Syndrome (SIRS)
MeSH Terms: conditions — Acute Lung Injury; Systemic Inflammatory Response Syndrome

ARMS (3):
- E1 (Experimental): This arm is conducted as a separate study (12-601-0001)
  Interventions: Drug: Sivelestat sodium hydrate
- E2 (Experimental): This arm is conducted as a separate study (12-603-0001).
  Interventions: Drug: Sivelestat sodium hydrate
- conventional therapy (No Intervention): This arm is conducted as a separate study (12-602-0001)

INTERVENTIONS:
Drug: Sivelestat sodium hydrate — 0.2 mg/kg/hr continuous i.v. infusion - up to 14 days
  Arms: E1
Drug: Sivelestat sodium hydrate — 0.2 mg/kg/hr continuous i.v. infusion - up to 14 days
  Arms: E2

SUMMARY:
The purpose of this study is to confirm the efficacy and safety of sivelestat in patients with acute lung injury associated with systemic inflammatory response syndrome. The results will be compared to the study with conventional treatment without sivelestat.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with systemic inflammatory response syndrome (SIRS)
2. Patients with acute lung injury (ALI) assessed using the criteria specified by the American-European Consensus Conference
3. Within 72 hours of onset of lung injury
4. Other inclusion criteria as specified in the protocol

Exclusion Criteria:

1. Already administrated Sivelestat before enrollment in the study
2. Neuromuscular disease that impairs spontaneous ventilation
3. Severe central nervous system disease
4. Bone marrow transplant
5. Lung transplant
6. Severe chronic liver disease
7. Neutropenia (neutrophil count: below 1000/mm3)
8. Other exclusion criteria as specified in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 649 (Actual)
Dates: Start 2004-06; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Ventilator free days (VFD) | 28 days

SECONDARY OUTCOMES:
28-day period survival rate, weaning rate from mechanical ventilation, intensive care unit (ICU) discharge rate, lung injury scores | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Development Planning, Study Director — Ono Pharmaceutical Co. Ltd
Locations (9):
- Japan (9):
  - Chugoku Region Facility, Chugoku
  - Chubu Region Facility, Chūbu
  - Hokkaido Region Facility, Hokkaido
  - Hokuriku Regional Facility, Hokuriku
  - Kanto Regional Facility, Kanto
  - Kinki Region Facility, Kinki
  - Kyushu Region Facility, Kyushu
  - Shikoku Region Facility, Shikoku
  - Tohoku Region Facility, Tōhoku